CLINICAL TRIAL: NCT00037817
Title: Phase I Study of Gene Induction Mediated by Sequential Decitabine/Depsipeptide Infusion With or Without Concurrent Celecoxib in Subjects With Pulmonary and Pleural Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020205; 02-C-0205; NCT00041158 (obsolete NCT alias)
Record Dates: First submitted 2002-05-21; First posted 2002-05-22 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2016-11-30

CONDITIONS: Advanced Esophageal Cancers; Primary Small Cell Lung Cancers; Non-Small-Cell Lung Carcinoma; Pleural Mesotheliomas; Cancers of Non-thoracic Origin With Metastases to the Lungs or Pleura
Keywords: Toxicity Evaluation; Pharmacokinetics; Apoptosis; Gene Induction; Gene Expression; Lung Cancer; Small Cell Lung Cancer; Non-Small Cell Lung Cancer; Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Small Cell Lung Carcinoma; Mesothelioma, Malignant | interventions — Decitabine; Depsipeptides; Celecoxib

ARMS (3):
- 1 (Experimental): Dose escalation cohort
  Interventions: Drug: Decitabine; Biological: Depsipeptide
- 2 (Experimental): Molecular response cohort
  Interventions: Drug: Decitabine; Biological: Depsipeptide
- 3 (Experimental): Celecoxib combination cohort at MTD
  Interventions: Drug: Decitabine; Biological: Depsipeptide; Drug: Celecoxib

INTERVENTIONS:
Drug: Decitabine — assigned dose level on day 4 and day 10 of each 34 day cycle
Biological: Depsipeptide — assigned dose level on day 4 and day 10 of each 34 day cycle
Drug: Celecoxib — 400mg PO BID on days 4 through 34 of each cycle
  Arms: 3

SUMMARY:
Background:

Previously we have demonstrated induction of tumor antigen and tumor suppressor gene expression in lung cancer cells following exposure to the DNA demethylating agent, Decitabine (DAC). We have also demonstrated that DAC mediated target gene expression and apoptosis can be significantly enhanced in cancer cells by subsequent exposure to the histone deacetylase (HDAC) inhibitor Depsipeptide FK228 (DP). Furthermore, we have demonstrated that following DAC, or DAC/DP exposure, cancer cells can be recognized by cytolytic T cells specific for the cancer testis antigen, NY-FSO-1.

This Phase I study will evaluate gene induction in thoracic oncology patients mediated by sequential DAC/DP treatment with or without the selective COX-2 inhibitor, celecoxib.

Objectives:

Evaluation of the pharmacokinetics and toxicity of continuous 72-hour intravenous Decitabine (DAC) infusion followed by 4-hour intravenous infusion of Depsipeptide FK228 (DP) with or without oral celecoxib in patients with unresectable cancers involving the lungs or pleura.

Analysis of NY-ESO-1, p16 and p21 expression in cancer specimens before and after sequential Decitabine/Depsipeptide treatment.

Analysis of serologic response to NY-ESO-1 before and after sequential drug treatment.

Analysis of apoptosis in tumor biopsies before and after sequential Decitabine/Depsipeptide treatment.

Refinement of laser capture microdissection and micro-array techniques for analysis of gene expression profiles in tumor tissues.

Eligibility:

Patients with histologically or cytologically proven primary small cell or non-small cell lung cancers, advanced esophageal cancers, pleural mesotheliomas, or non-thoracic cancers with metastases to the lungs or pleura.

Patients must be 18 years or older with an ECOG performance status of 0-2 and have adequate pulmonary reserve evidenced by FEV1 and DLCO greater than the 30% predicted, and less than 50 mm Hg and p02 greater than 60 mm Hg on room air ABG.

Patients must have a platelet count greater than 100.000. an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of less than 1.5 x upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

Design:

Patients with inoperable malignancies involving lungs or pleura will receive two cycles of 72-hour intravenous infusion of Decitabine followed by 4-hour Depsipeptide infusion using a Phase I study design.

Decitabine will be administered by continuous infusion on days 1-4, and patient cohorts will receive escalating doses of Depsipeptide administered on day 4 and day 10 of a 34 day cycle.

Once the MTD and toxicities for sequential DAC/DP have been identified, additional cohorts of 6 lung cancer patients and 6 mesothelioma patients will receive sequential DAC/DP administered at the MTD as outlined above with celecoxib (400mg bid) administered on days 4-34 of each treatment cycle, as a means to enhance target cell apoptosis and facilitate anti-tumor immune recognition/response.

Pharmacokinetics, systemic toxicity, and response to therapy will be recorded. Tumor biopsies will be obtained prior to, and after therapy to evaluate expression of NY-ESO-1 tumor antigen, as well as p16 and p21 tumor suppressor genes, which are known to be modulated by chromatin structure. Additional analysis will be undertaken to evaluate the extent of apoptosis in tumor tissues, and to determine if immune recognition of NY-ESO-1 can be demonstrated following sequential DAC?DP +/- celecoxib treatment.

As the exact set of comparisons and analyses to be performed will be determined following completion of the trial and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.

A total of 40 patients will be enrolled.

DETAILED DESCRIPTION:
Background:

Previously we have demonstrated induction of tumor antigen and tumor suppressor gene expression in lung cancer cells following exposure to the DNA demethylating agent, Decitabine (DAC). We have also demonstrated that DAC mediated target gene expression and apoptosis can be significantly enhanced in cancer cells by subsequent exposure to the histone deacetylase (HDAC) inhibitor Depsipeptide FK228 (DP). Furthermore, we have demonstrated that following DAC, or DAC/DP exposure, cancer cells can be recognized by cytolytic T cells specific for the cancer testis antigen, NY-FSO-1.

This Phase I study will evaluate gene induction in thoracic oncology patients mediated by sequential DAC/DP treatment with or without the selective COX-2 inhibitor, celecoxib.

Objectives:

Evaluation of the pharmacokinetics and toxicity of continuous 72-hour intravenous Decitabine (DAC) infusion followed by 4-hour intravenous infusion of Depsipeptide FK228 (DP) with or without oral celecoxib in patients with unresectable cancers involving the lungs or pleura.

Analysis of NY-ESO-1, p16 and p21 expression in cancer specimens before and after sequential Decitabine/Depsipeptide treatment.

Analysis of serologic response to NY-ESO-1 before and after sequential drug treatment.

Analysis of apoptosis in tumor biopsies before and after sequential Decitabine/Depsipeptide treatment.

Refinement of laser capture microdissection and micro-array techniques for analysis of gene expression profiles in tumor tissues.

Eligibility:

Patients with histologically or cytologically proven primary small cell or non-small cell lung cancers, advanced esophageal cancers, pleural mesotheliomas, or non-thoracic cancers with metastases to the lungs or pleura.

Patients must be 18 years or older with an ECOG performance status of 0-2 and have adequate pulmonary reserve evidenced by FEV1 and DLCO greater than the 30% predicted, and less than 50 mm Hg and p02 greater than 60 mm Hg on room air ABG.

Patients must have a platelet count greater than 100.000. an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of less than 1.5 x upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

Design:

Patients with inoperable malignancies involving lungs or pleura will receive two cycles of 72-hour intravenous infusion of Decitabine followed by 4-hour Depsipeptide infusion using a Phase I study design.

Decitabine will be administered by continuous infusion on days 1-4, and patient cohorts will receive escalating doses of Depsipeptide administered on day 4 and day 10 of a 34 day cycle.

Once the MTD and toxicities for sequential DAC/DP have been identified, additional cohorts of 6 lung cancer patients and 6 mesothelioma patients will receive sequential DAC/DP administered at the MTD as outlined above with celecoxib (400mg bid) administered on days 4-34 of each treatment cycle, as a means to enhance target cell apoptosis and facilitate anti-tumor immune recognition/response.

Pharmacokinetics, systemic toxicity, and response to therapy will be recorded. Tumor biopsies will be obtained prior to, and after therapy to evaluate expression of NY-ESO-1 tumor antigen, as well as p16 and p21 tumor suppressor genes, which are known to be modulated by chromatin structure. Additional analysis will be undertaken to evaluate the extent of apoptosis in tumor tissues, and to determine if immune recognition of NY-ESO-1 can be demonstrated following sequential DAC?DP +/- celecoxib treatment.

As the exact set of comparisons and analyses to be performed will be determined following completion of the trial and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.

A total of 40 patients will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically or cytologically proven primary small cell or non-small cell lung cancers, advanced esophageal cancer, or pleural mesotheliomas are eligible for evaluation. In addition, patients with cancers of nonthoracic origin with metastases to the lungs or pleura are eligible for evaluation.

Patients with intracranial metastases which have been treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids following treatment.

Patients with prior Decitabine or Depsipeptide exposure are eligible for study provided they have not experienced dose limiting toxicity at the dose of DAC or DP that they are scheduled to receive.

Patients with prior or current celecoxib exposure are eligible for study provided that it has been intermittent, or of short term duration (less than 1 month).

Patients must have had no chemotherapy, biologic therapy, celecoxib exposure, or radiation therapy for their malignancy within 30 days prior to treatment. Patients may have received localized radiation therapy to non-target lesions provided that the radiotherapy is completed 14 days prior to commencing therapy, and the patients has recovered from any toxicity.

Patients must have an ECOG performance status of 0-2.

Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO greater than the 30% predicted, and pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG.

Patients must be 18 years of age or older due to the unknown effects of demethylating agents and HDAC inhibitors during childhood and adolescent development.

Patients must have a platelet count greater than 100, 000, an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of less than 1.5 x upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

All patients will have cardiology consultation. Subsequent evaluation will consist of stress/redistribution thallium, 24th ambulatory EKG monitoring, ECHO, cardiac MR, or coronary angiography as indicated.

Patients must be aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks. The patient must be willing to sign an informed consent, and undergo tumor biopsies to evaluate target gene expression prior to, and after, decitabine/depsipeptide treatment.

EXCLUSION CRITERIA:

Patients with primary and metastatic cancers involving the lungs or pleura which cannot be readily biopsied by endoscopic or percutaneous fine needle aspiration techniques will be excluded.

Patients with untreated limited stage SCLC, and operable NSCLC or operable esophageal cancer will be excluded.

Patients who have received three or more systemic cytotoxic treatment regimens will be excluded due to possible cumulative marrow suppression.

Patients with active intracranial and leptomeningeal metastases as well as those requiring anticonvulsant medications will be excluded.

Patients with life expectancy less than three months will be excluded.

Patients with pulmonary embolism, or deep venous thrombosis, or prosthetic heart valves requiring anticoagulation will be excluded.

Cardiac exclusion criteria, patients with known cardiac abnormalities such as:

-Uncontrolled arrhythmias

History of serious ventricular arrhythmias not controlled by coronary artery bypass surgery.

Patients with a history of sustained VT, VF, Toursades de Pointes, or cardiac arrest who do not have an automatic implantable cardioverter defibrillator in place

Congenital Long QT syndrome or QTc greater than 480 msec

Patients with Mobitz II second degree block who do not have a pacemaker

Patients with any cardiac arrhythmia requiring anti-arrhythmic medication other than a beta blocker or calcium channel blocker

Patients in whom digitalis cannot be discontinued

* Decompensated heart failure (NYHA Class II or IV)
* LVEF less than 50% by MUGA scan or echocardiogram
* Hypertrophic or restrictive cardiomyopathy from prior treatment of other causes and patients with left ventricular hypertrophy
* Uncontrolled hypertension (i.e greater than or equal to 160/95)
* Myocardial infarction within one year of study
* Clinical significant active myocardial ischemia on the basis of nuclear imaging or angiography
* History of coronary artery disease (e.g. angina Canadian Class II-Iv or positive stress imaging study)
* Patients with other cardiac disease may be excluded at the discretion of the PI following consultation with cardiology

Co-medication causing QTc prolongation unless a 5 half-life washout period has elapsed between discontinuing the drug and entering this study.

Pregnant patients and lactating mothers will be excluded due to the unknown, potentially harmful effects of demethylating agents and HDAC inhibitors on fetal and early childhood development.

Patients with active infections will be excluded.

Patients with HIV infection will be excluded due to the potential risk of opportunistic infection during DAC/DP-induced myelosuppression and potentially deleterious activation of viral gene expression.

Patients should not be using hydrochlorothiazide diuretics if entered on this protocol. Therefore, patients who must use hydrochlorothiazide diuretics will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2002-05-17; Primary Completion 2008-10-08 (Actual); Study Completion 2009-11-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics and toxicity profile | Every cycle until approximately 70 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schrump DS, Nguyen DM. Targets for molecular intervention in multistep pulmonary carcinogenesis. World J Surg. 2001 Feb;25(2):174-83. doi: 10.1007/s002680020016. PMID 11338019
- [Background] Schrump DS, Waheed I. Strategies to circumvent SV40 oncoprotein expression in malignant pleural mesotheliomas. Semin Cancer Biol. 2001 Feb;11(1):73-80. doi: 10.1006/scbi.2000.0348. PMID 11243901
- [Background] Baylin SB, Esteller M, Rountree MR, Bachman KE, Schuebel K, Herman JG. Aberrant patterns of DNA methylation, chromatin formation and gene expression in cancer. Hum Mol Genet. 2001 Apr;10(7):687-92. doi: 10.1093/hmg/10.7.687. PMID 11257100